CLINICAL TRIAL: NCT01719952
Title: Comparison of Haemodynamic and Cardiovascular Effects of Carbetocin and Oxytocin in Women Undergoing Elective Caesarean Section: A Double-blinded Randomised Clinical Trial
Brief Title: Haemodynamic and Cardiovascular Effects of Carbetocin and Oxytocin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Nirmala Chandralega Kampan, MRCOG(UK), Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKMMC
Record Dates: First submitted 2012-07-06; First posted 2012-11-01 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Pregnancy Related; Anaesthesia
Keywords: pregnancy; anaesthesia; caesarean section
MeSH Terms: interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbetocin (Experimental): Carbetocin 100 µg, given as an intravenous bolus over 30 seconds others names are: duratocin, pabal
  Interventions: Drug: Carbetocin
- Oxytocin (Active Comparator): Other names are Pitocin, syntocinon given as an intravenous bolus over 30 seconds by the anaesthetist following clamping of the umbilical cord only in patient that has been randomized to this group.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — IV carbetocin 100mcg, only in selected patient given as an intravenous bolus over 30 seconds by the anaesthetist following clamping of the umbilical cord only in patient that has been randomized to this group.
  pitocin 5 IU also given as an intravenous bolus over 30 seconds by the anaesthetist following clamping of the umbilical cord only in patient that has been randomized to this group.
  Other Names: Duratocin for carbetocin; pitocin for oxytocin
  Arms: Carbetocin
Drug: Oxytocin — 5 IU given as an intravenous bolus over 30 seconds by the anaesthetist following clamping of the umbilical cord only in patient that has been randomized to this group.
  Other Names: pitocin
  Arms: Oxytocin

SUMMARY:
A double-blinded randomised control trial conducted in the Department of Obstetrics and Gynaecology of a tertiary hospital, Universiti Kebangsaan Malaysia Medical Centre (UKMMC) for two years duration from January 1st, 2012 till December 31st, 2013.

The aim of the study is to compare the haemodynamic and cardiovascular effects between intravenous carbetocin 100 μg and intravenous oxytocin 5 IU in women undergoing elective Lower Segment Caesarean Section (EL LSCS).

Study hypothesis: A single injection of carbetocin is haemodynamically and cardiovascularly safe and has similar efficacy in comparison to a single injection of oxytocin.

DETAILED DESCRIPTION:
OUTCOME MEASURES systolic blood pressure (SBP), diastolic blood pressure (DBP), Heart Rate (HR), saturation of oxygen (SpO2) in certain time after drug injection.

The presence of myocardial ischemia symptoms and side effects of both drugs, ECG changes such as ST depression and changes in T-waves.

Hemoglobin and troponin-T level

The need for additional oxytocin infusion and estimated blood loss

The time interval between initial drug administration, type of additional oxytocic intervention that used and complication that happened.

ELIGIBILITY:
Inclusion Criteria:

1. Viable, singleton pregnancy ≥ 37 weeks gestation undergoing EL LSCS.
2. Low risk for post-partum hemorrhage, such as no proven abruptio placentae, placenta previa, multiple pregnancy, pre-eclampsia / gestational hypertension, previous PPH, obesity (based on BMI pre pregnancy which is ≥ 30 kg/m2), big baby.
3. Ability to provide informed consent.

Exclusion Criteria:

1. Emergency caesarean section
2. Preterm Labour
3. Grandmultipara
4. Multiple Pregnancy
5. Placenta Previa
6. Previous PPH
7. Maternal Obesity ( BMI pre pregnancy ≥ 30 kg/m2))
8. Have co-morbidity illness such as hypertension/pre-eclampsia, established cardiac diseases, history or evidence of liver, renal, vascular, or endocrine disease and bleeding disorder.
9. Contraindication to carbetocin and oxytocin
10. Language Barrier
11. Women undergoing general anaesthesia
12. Women who has abnormal baseline ECG that suggestive myocardial ischemia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Haemodynamic effects | 2 years
  1. Haemodynamic effect (blood pressure, heart rate, saturation of oxygen)
  2. Presence of ECG changes such as ST depression and changes in T-waves
  3. Presence of myocardial ischemia symptoms (such as chest pain, shortness of breath, feeling of heaviness in chest pain)
  4. To compare the troponin T levels

SECONDARY OUTCOMES:
Blood loss measurement | 2 years
  1. Need for additional oxytocin infusion
  2. Total blood loss
  3. Drop in haemoglobin level post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Nirmala C Kampan, MRCOG(UK), Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Department of O&G, Cheras, Kuala Lumpur, Malaysia